CLINICAL TRIAL: NCT05118620
Title: Pericapsular Nerve Group Block (PENG): A Randomized, Triple-Masked, Placebo-Controlled Clinical Trial
Brief Title: Pericapsular Nerve Group Block (PENG) for Hip Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of staff to enroll
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PENG Block for Hip Surgery
Record Dates: First submitted 2021-10-20; First posted 2021-11-12 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Hip Arthropathy; Postoperative Pain, Acute; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Care Provider, Investigators/Outcomes Assessors) Study solution containing either local anesthetic (bupivacaine) or normal saline will be prepared by the University of California San Diego Investigational Drug Study Service. Both bupivacaine and normal saline are clear and indistinguishable visually.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active Treatment (Experimental): This group will receive a single injection PENG nerve block of bupivacaine 0.375% (20 mL)
  Interventions: Drug: Active bupivacaine 0.375% PENG block
- Placebo (Placebo Comparator): This group will receive a single injection PENG nerve block with normal saline (20 mL)
  Interventions: Drug: Placebo normal saline PENG block

INTERVENTIONS:
Drug: Active bupivacaine 0.375% PENG block — A PENG block with bupivacaine 0.375% and epinephrine will be administered using ultrasound-guidance
  Other Names: Active Pericapsular Nerve Group block
  Arms: Active Treatment
Drug: Placebo normal saline PENG block — A PENG block with normal saline and epinephrine will be administered using ultrasound-guidance
  Other Names: Placebo Pericapsular Nerve Group block
  Arms: Placebo

SUMMARY:
This will be a randomized comparison of pericapsular nerve group (PENG) blocks with bupivacaine and a placebo control (PENG blocks with normal saline). The overall objective of the proposed research is to determine the relative risks and benefits of a single-injection PENG block to provide postoperative analgesia following hip arthroscopy.

Hypothesis 1: Following hip arthroscopy, participants with a PENG block will experience less pain in the recovery room compared with current standard-of-care as measured with the Numeric Rating Scale (NRS).

Hypothesis 2: Following hip arthroscopy, participants with a PENG block will consume less opioid in the operating and recovery rooms compared with current standard-of-care as measured in oral morphine milligram equivalents.

Primary end point: In order to claim that PENG blocks are superior to placebo overall, at least one of these two hypotheses must demonstrate PENG superiority while the other cannot demonstrate inferiority.

DETAILED DESCRIPTION:
Following painful surgical procedures of the hip, postoperative analgesia is often provided simply with intravenous and oral analgesics. Peripheral nerve blocks using local anesthetic have been investigated, and while they do provide analgesia, they all carry a high risk of inducing weakness of the quadriceps and/or hip adductors. This, in turn, results in an unacceptably high risk of subsequent falls, and peripheral nerve blocks are therefore not standard-of-care at most health centers. For example, at the University of California San Diego hospitals, no peripheral nerve block is provided even for the most painful hip surgery, hip arthroplasty. This results in a strong dependence on opioid analgesics which frequently provide inadequate analgesia and have undesirable side effects for both individuals and society. Peripheral nerve blocks with local anesthetic can provide analgesia for over 12 hours without any systemic side effects. Thus, it would be preferable to provide peripheral nerve blocks to patients having painful hip surgery to reduce pain as well as decrease opioid use and their associated adverse side effects. Recently, a new type of block has been reported to provide analgesia to the hip joint: the "pericapsular nerve group" (PENG) block. Twenty case reports and series have been published suggesting potent analgesia while not inducing any motor block. However, no randomized, controlled clinical trial is available to validate the technique and quantify both risks and benefits. The investigators therefore propose such a study.

This investigation will be a randomized, triple-masked, placebo-controlled, parallel-arm, human subjects clinical trial. Adults undergoing painful unilateral primary hip arthroscopy with general anesthesia will be offered enrollment. Of note, the investigators will be using standard-of-care analgesics including oral and intravenous opioids as well as surgeon-infiltrated local anesthetic directly into the wound under an FDA-approved purpose and do not plan to research a possible change of indication or use of these medications as part of this research project. These treatments will be administered in both groups constituting our institution standard-of-care.

Following written, informed consent, all participants will have a peripheral intravenous catheter inserted and standard noninvasive monitors applied. The investigators will evaluate muscle strength with an isometric force electromechanical dynamometer (MicroFET2, Lafayette Instrument Company, Lafayette, IN) to measure the force produced during a maximum voluntary isometric contraction (MVIC) in a seated position with the knees flexed at 90º. For quadriceps femoris evaluation, the dynamometer will be placed on the ipsilateral anterior tibia perpendicular to the tibial crest just proximal to the medial malleolus. For hip adductor evaluation, the femoral shaft will be held at 30º off midline and the dynamometer placed over the medial femoral epicondyle (adductor tubercle). For all measurements, participants will be asked to take 2 seconds to come to maximum effort contracting the target muscle(s), maintain this effort for 5 sec, and then relax. The measurements immediately prior to perineural ropivacaine administration will be designated baseline measurements, and all subsequent measurements will be expressed as a percentage of the pre-infusion baseline. Participants who cannot perform these maneuvers will have their data excluded from the muscle strength calculations (i.e., a "zero" will not be entered for these participants).

Participants will then be randomized using a computer-generated list to one of two treatment groups (blocks of 4): a PENG block with 20 mL of either (1) bupivacaine 0.375% or (2) normal saline [epinephrine added to both]. Investigational pharmacists will create the lists and fill syringes with one of the two possible study solutions and provide investigators with syringes that will not identify the treatment. Bupivacaine and normal saline are identical in appearance, and all investigations, patients, and clinical staff will remain masked to treatment group. Following enrollment completion, the Investigational Drug Service will provide the statistician with lists of the treatment groups labeled "A" and "B". Only following statistical analysis will the specific treatment groups be identified by the Investigational Drug Service so that the investigators may prepare the manuscript reporting the results (termed "triple masked").

All blocks will be placed by a regional anesthesia fellow or resident under the direct supervision and guidance of a regional anesthesia attending (or by the attending themselves). Participants will have supplemental oxygen administered via a nasal cannula or face mask and placed in the supine position. Intravenous midazolam and fentanyl will be titrated for patient comfort, while ensuring that patients remain responsive to verbal cues.

Blocks technique: A low-frequency curved-array ultrasound transducer will be placed in a transverse plane over the anterior inferior iliac spine "and then aligned with the pubic ramus by rotating the probe counterclockwise approximately 45 degrees. In this view the iliopubic eminence, the iliopsoas muscle and tendon, the femoral artery, and pectineus muscle" are observed. A 17-gauge needle will be inserted using an in-plane technique directed medially. The needle tip will be inserted in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly. After gentle negative aspiration, the study fluid will be slowly injected with frequent aspiration.

Twenty to 30 minutes following the initial local anesthetic bolus injection, muscle strength will be evaluated and recorded in the same manner as the baseline measurements.

Intraoperatively, all participants will receive a general anesthetic using inhaled and intravenous anesthetic and oxygen. Intravenous fentanyl and/or morphine will be administered for cardiovascular responsiveness to noxious stimuli at the discretion of the anesthesia provider.

Postoperatively, participants will be discharged with a prescription for oxycodone 5 mg tablets for supplementary analgesia and instructed to record the time at which they take their first opioid tablet as well as the time at which they believe the block starts to wear off. If a study subject is admitted to the hospital, the investigators will continue to follow as described herein.

Outcome measurements. Within the recovery room, pain scores, opioid requirements, and antiemetic administration will be recorded by nursing staff masked to treatment group assignment. The morning following surgery, all participants will be contacted by phone or in person [if hospitalized] to record outcomes. For outpatients, opioid requirements will be recorded during the call, while inpatients will have opioid requirements extracted from the electronic medical record. In addition, the investigators will extract antiemetic use from the electronic record.

Analysis Plan:

In order to claim that PENG blocks are superior to placebo overall, at least one of these two hypotheses must demonstrate PENG superiority while the other cannot demonstrate inferiority:

Hypothesis 1: Following hip arthroscopy, participants with a PENG block will experience less pain in the recovery room compared with current standard-of-care as measured with the Numeric Rating Scale (NRS).

Hypothesis 2: Following hip arthroscopy, participants with a PENG block will consume less opioid in the operating and recovery rooms compared with current standard-of-care as measured in oral morphine milligram equivalents.

Secondary hypotheses are as follows (postoperative day 1 data collection for all):

Hypothesis 2.1: Average and worst pain with movement Hypothesis 2.2: Opioid consumption; average and worst pain at rest Hypothesis 2.3: Awakenings due to pain and difficulty sleeping due to pain

Primary test will be for superiority of bupivacaine over saline. If tests of superiority fail, exploratory tests for noninferiority will follow with margins specified.

Baseline characteristics of the randomized groups will be summarized with means, standard deviations, and quartiles. Balance between groups will be assessed. Specifically, standardized differences will be calculated using Cohen's d whereby the difference in means or proportions is divided by the pooled standard deviation estimates. Any key variables (age, sex, height, weight, and BMI) with an absolute standardized difference >1.96 x square root of 2/n, where n is the sample size per group will be noted and included in a linear regression model to obtain an estimate of the treatment group differences adjusted for the imbalanced covariate(s). If residuals from the linear regression indicate violations of key assumptions (i.e. homoscedasticity or Gaussian distribution), data transformations and/or alternative generalized linear models will be applied as appropriate. If all key covariates are found to be balanced between groups, the Wilcoxon-Mann-Whitney test will be used for primary inference. Secondary outcomes will also be analyzed by Wilcoxon-Mann-Whitney test, or linear models (or generalized linear models) as appropriate to adjust for any imbalanced covariates.

Family-wise Error Control. Hypotheses will be tested with strong control of the family-wise error rate at 5%. Testing begins with equally weighted co-primary hypotheses H11 and H12. If either of these are significant at the 0.05/2 = 0.025 level, that alpha is passed on to other hypotheses following the arrows in the figure. For example, if the p-value for H12 is less than 0.025, but the p-value for H11 is not, then H11 can be tested at the 0.025 + 0.025/2 = 0.0375 level. If both H11 and H12 are rejected, no alpha is spent, and the investigators go on to similarly test H21a, H21b, H22a, H22b, and H23a, and H23b. If a given test does not reach local significance, alpha is spent and cannot be passed along to hypotheses further along the graph.

Sample size justification. Simulated Power for NRS: Simulated Power for NRS. YaDeau et al. (2012) reports mean +/- standard deviation NRS pain score at rest of 4.2 +/- 1.8 NRS units. The investigators simulated data from the distribution shown in Figure below, which yields mean standard deviation of 4.2 +/- 1.8 and 3.0 +/- 1.7. Based on 1,000 simulated trials the investigators found a sample size of n=50 per group provides 85.7% power with two-sided alpha =2.5%.

YaDeau (2012) reports mean +/- standard deviation NRS pain score with movement (0-10) at 24 hours of 5.5 +/- 2.3 NRS units. The investigators simulated data from the distribution, which yields mean +/- standard deviation of 5.5 2.6 and 3.9 +/- 2.5. Based on 1,000 simulated trials the investigators found a sample size of n=50 per group provides 83% power with two-sided alpha=2.5%.

Simulated Power for opioid consumption. Opioid consumption was assumed to follow a truncated normal distribution with mean 29 +/- 21 mg (as reported in YaDeau et al. (2012)). A sample size of n = 50 per group provides about 84% power to detect a treatment difference as small as 18 mg (mean of 29 mg with normal saline vs 11 mg with bupivacaine) with two-sided alpha = 2.5%.

Therefore, the investigators will enroll 50 participants for each of two treatments with primary end point values for a total enrollment of 100 participants. To allow for dropouts, the investigators request a maximum enrollment of 120 participants.

ELIGIBILITY:
Inclusion Criteria:

* undergoing unilateral primary hip arthroscopy with at least moderate postoperative pain anticipated
* analgesic plan includes a general anesthetic
* age 18 years or older

Exclusion Criteria:

* morbid obesity as defined by a body mass index > 40 (BMI=weight in kg / [height in meters]2)
* any planned regional analgesic or anesthetic
* chronic opioid use (daily use within the 2 weeks prior to surgery and duration of use > 4 weeks)
* history of opioid abuse
* any comorbidity which results in moderate or severe functional limitation
* inability to communicate with the investigators or hospital staff
* pregnancy
* incarceration
* any reason for increased risk of a peripheral nerve block (e.g. anticoagulation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Pain scores within the recovery room as measured using the numeric rating scale, collected postoperative day 1 for the time since midnight. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale | From admission to the recovery room following surgery until discharge from the recovery room, assessed up to 72 hours. In order to claim PENG blocks are superior to placebo overall at least 1 of the 2 primary hypotheses must demonstrate PENG superiority
  Pain measured using the numeric rating scale, collected within the recovery room for the time since midnight. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain
Total opioid consumption within the recovery room (measured in intravenous morphine equivalents) | From admission to the recovery room following surgery until discharge from the recovery room, assessed up to 72 hours. In order to claim PENG blocks are superior to placebo overall at least 1 of the 2 primary hypotheses must demonstrate PENG superiority
  Total opioid consumption within the recovery room (measured in intravenous morphine equivalents)

SECONDARY OUTCOMES:
"Average" pain with movement during postoperative day 1 as measured using the numeric rating scale, collected postoperative day 1. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale | From discharge from the recovery room until the data collection phone call on postoperative day 1
  "Average" pain with movement during postoperative day 1 as measured using the numeric rating scale, collected postoperative day 1 for the time since discharge from the recovery room. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale
"Worst" pain with movement on postoperative day 1 as measured using the numeric rating scale, collected postoperative day 1. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale | From discharge from the recovery room until the data collection phone call on postoperative day 1
  "Worst" pain during postoperative day 1 as measured using the numeric rating scale, collected postoperative day 1 for the time since discharge from the recovery room. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale
"Average" pain at rest on postoperative day 1 as measured using the numeric rating scale, collected postoperative day 1. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale | From discharge from the recovery room until the data collection phone call on postoperative day 1
  "Average" pain at rest on postoperative day 1 as measured using the numeric rating scale, collected postoperative day 1 for the time since discharge from the recovery room. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale
"Worst" pain at rest on postoperative day 1 as measured using the numeric rating scale, collected postoperative day 1. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale | From discharge from the recovery room until the data collection phone call on postoperative day 1
  "Worst" pain at rest on postoperative day 1 as measured using the numeric rating scale, collected postoperative day 1 for the time since discharge from the recovery room. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale
Total opioid consumption from recovery room discharge until the data collection phone call on postoperative day 1(measured in intravenous morphine equivalents) | From recovery room discharge until the data collection phone call on postoperative day 1
  Total opioid consumption from recovery room discharge until the data collection phone call on postoperative day 1(measured in intravenous morphine equivalents)
Difficulty sleeping due to pain the evening of surgery | Difficulty sleeping due to pain the evening of surgery, assessed the day following surgery
  Difficulty sleeping due to pain the evening of surgery as either "yes" or "no", assessed the day following surgery
Awakenings to pain the evening of surgery | The number of awakenings due to pain the evening of surgery, assessed the day following surgery
  The number of awakenings due to pain the evening of surgery, assessed the day following surgery
Change in quadriceps strength between pre- and post-block measurements, as measured with an isometric force electromechanical dynamometer | Immediately before and 20-30 minutes after application of the nerve block
  Change in maximum voluntary isometric contraction of the quadriceps muscle between pre- and post-block measurements, as measured with an isometric force electromechanical dynamometer. For quadriceps femoris evaluation, the dynamometer will be placed on the ipsilateral anterior tibia perpendicular to the tibial crest just proximal to the medial malleolus. For all measurements, participants will be asked to take 2 seconds to come to maximum effort contracting the target muscle(s), maintain this effort for 5 sec, and then relax. The measurements immediately prior to perineural ropivacaine administration will be designated baseline measurements, and all subsequent measurements will be expressed as a percentage of the pre-infusion baseline.
Change in hip adductor strength between pre- and post-block measurements, as measured with an isometric force electromechanical dynamometer | Immediately before and 20-30 minutes after application of the nerve block
  Change in maximum voluntary isometric contraction of the hip adductors between pre- and post-block measurements, as measured with an isometric force electromechanical dynamometer. For hip adductor evaluation, the femoral shaft will be held at 30º off midline and the dynamometer placed over the medial femoral epicondyle (adductor tubercle). For all measurements, participants will be asked to take 2 seconds to come to maximum effort contracting the target muscle(s), maintain this effort for 5 sec, and then relax. The measurements immediately prior to perineural ropivacaine administration will be designated baseline measurements, and all subsequent measurements will be expressed as a percentage of the pre-infusion baseline.

OTHER OUTCOMES:
Time to perform peripheral nerve block, as measured from the time the needle first touches the patient until it is withdrawn for the final time. | Preoperatively
  Time to perform peripheral nerve block, as measured from the time the needle first touches the patient until it is withdrawn for the final time.
Study fluid injection time as measured in military format | Preoperatively
  The time at which the study fluid is injected for the PENG block
"Lowest" pain at rest on postoperative day 1 as measured using the numeric rating scale, collected postoperative day 1. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale | From discharge from the recovery room until the data collection phone call on postoperative day 1
  "Lowest" pain at rest on postoperative day 1 as measured using the numeric rating scale, collected postoperative day 1 for the time since discharge from the recovery room. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale
"Current" pain at rest on postoperative day 1 as measured using the numeric rating scale, collected postoperative day 1. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale | At the time of the data collection phone call on postoperative day 1
  "Current" pain at rest on postoperative day 1 as measured using the numeric rating scale, collected postoperative day 1. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale
Number of falls from the time of recovery room discharge until the data collection phone call on postoperative day 1 | From recovery room discharge until the data collection phone call on postoperative day 1
  The number of falls from the time of recovery room discharge until the data collection phone call on postoperative day 1
Cumulative opioid consumption postoperative day 1 (measured in oral oxycodone equivalents) | From recovery room discharge until the data collection phone call on postoperative day 1
  Cumulative opioid consumption postoperative day 1 (measured in oral oxycodone equivalents)
Subjective weakness in the hip joint | At the time of the data collection phone call on postoperative day 1
  If the participant feels that they have weakness of the muscles that innervate the hip (binary answer of "yes" or "no")
Time of first opioid use following recovery room discharge recorded in military time format | From recovery room discharge until the data collection phone call on postoperative day 1
  Time of first opioid use following recovery room discharge recorded in military time format
Time of block resolution (subjective) recorded in military time format | From recovery room discharge until the data collection phone call on postoperative day 1
  Time of first opioid useTime of block resolution (subjective) recorded in military time format following recovery room discharge recorded in military time format
Total opioid consumption within the operating room (measured in intravenous morphine equivalents) | From arrival in the operating room until operating room discharge to the recovery room, assessed for up to 72 hours
  The total number of milligrams of opioid consumption within the operating room (measured in intravenous morphine equivalents)
Anti-emetic consumption within the recovery room | From admission to the recovery room until discharge from the recovery room, assessed for up to 72 hours
  Anti-emetic consumption within the recovery room as a binary variable ("yes" or "no")
Surgical start as recorded using military time format | During surgery
  The time of the surgical incision as recorded using military time format
Surgical stop as recorded using military time format | During surgery
  The time of the final suture insertion as recorded using military time format

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, MD, MS, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided